CLINICAL TRIAL: NCT04266080
Title: Assessing a Game-Based Physical Activity Intervention in Childhood Cancer Survivors: The STEP UP for FAMILIES Pilot Study
Brief Title: Game-Based Physical Activity in Childhood Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sohn Conference Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-040
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Survivors of Childhood Cancer
Keywords: Game-Based; Physical Activity; 20-040
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a single-arm pilot study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- childhood cancer survivors & and one parent/legal guardian (Experimental): The study plans to recruit 30 childhood cancer survivors and a parent/legal guardian for each survivor. Participants will be provided with a Fitbit Inspire HR wearable device to record their step counts for two weeks pre-intervention, and over the six-month follow-up period (3-month intervention and 3month follow-up).
  Interventions: Other: Fitbit Inspire HR; Other: Questionaires

INTERVENTIONS:
Other: Fitbit Inspire HR — assessing step counts
Other: Questionaires — Patient-Reported Outcomes Measurement Information System (PROMIS)

SUMMARY:
This study will test whether a game-based exercise plan can help increase the level of physical activity in childhood cancer survivors. The game-based exercise plan will involve participation by both a childhood cancer survivor and his/her parent or caregiver. This study will also look at whether the game-based exercise plan improves childhood cancer survivors' quality of life.

ELIGIBILITY:
Inclusion Criteria:

Childhood cancer survivor:

* History of treatment for childhood cancer with cardiotoxic therapy (anthracyclines, chest radiation, total body irradiation)
* Off all systemic cancer therapy for ≥ 2 years
* Ability to speak and understand English
* Ability to complete all protocol assessments
* Mobile device with SMS text messaging capability
* Ambulatory and able to perform all study requirements
* Attained age 10-16 years
* Has a parent or legal guardian willing to participate in the study as a dyad
* Willing to receive daily SMS text message alerts
* Not currently exercising at least 30 minutes per day (5 days/week)
* ECOG Performance Status of 0-1

Parent/legal guardian:

* Parent or legal guardian of a childhood cancer survivor treated with cardiotoxic therapy (anthracyclines, chest radiation, total body irradiation)
* Parent or legal guardian of a child age 10-16 years who is at least 2 years from completion of systemic cancer therapy
* Ability to speak and understand English
* Ability to complete all protocol assessments
* Ability to provide informed consent
* Ambulatory and able to perform all study requirements
* Access to a mobile device with SMS text messaging capability
* Is the parent or legal guardian of a childhood cancer survivor who is willing to participate in this study as a dyad
* Willing to receive daily SMS text message alerts
* ECOG Performance Status of 0-1

Exclusion Criteria:

* Survivors, or parents/legal guardians of survivors, with a medical condition that makes it unsafe to complete study requirements are not eligible for this study. This includes a diagnosis of:

  * Severe persistent asthma
  * Known symptomatic coronary artery disease
  * Musculoskeletal defects that interfere with sustained physical activity
  * Any medical or psychosocial condition that, in the opinion of the investigator, would jeopardize the health of the participant during study procedures

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention | 3 months
  (i.e., all four responses on the AIM rates as either a 4 or 5 on a 5-point Likert scale of acceptability);

SECONDARY OUTCOMES:
step count | 3 months
  step count by FitBit-type devices
hours of sleep per night | 3 months
  by FitBit-type devices

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Friedman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm